CLINICAL TRIAL: NCT00355069
Title: Better Pediatric Asthma Outcomes Through Chronic Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Judith Fifield, Professor & Director, Ethel Donaghue TRIPP Center, UConn Health
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1U18HS011068-01 (AHRQ); U18HS011068 (AHRQ)
Record Dates: First submitted 2006-07-19; First posted 2006-07-21 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Asthma
Keywords: pediatric; asthma; translational research; health information technology
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): Received the Basic Pediatric Chronic Care Model AND the Medication Assessment Prompt AND family education
  Interventions: Behavioral: electronic (computer based) provider feedback tool
- 2 (Experimental): Received the Basic Pediatric Chronic Care Model AND the Medication Assessment Prompt but NOT family education
  Interventions: Behavioral: electronic (computer based) provider feedback tool
- 3 (Experimental): Received the Basic Pediatric Chronic Care Model AND family education but NOT the Medication Assessment Prompt
  Interventions: Behavioral: electronic (computer based) provider feedback tool
- 4 (Placebo Comparator): Received the Basic Pediatric Chronic Care Model only (NO Medication Assessment Prompt and NO family education)
  Interventions: Behavioral: electronic (computer based) provider feedback tool

INTERVENTIONS:
Behavioral: electronic (computer based) provider feedback tool — All sites received a Basic Pediatric Chronic Care Model; 2x2 factorial design allocated the additional Medication Assessment Prompt and family education across the four sites as well.
  Other Names: UCAN Control Asthma Program; Medication Assessment Prompt (MAP)

SUMMARY:
This 3-year, multi-site study focuses on the translation of cost-effective methods to bring a chronic care model to the care of poor, minority, inner-city children with asthma, at risk of the worst outcomes for the leading chronic disease of children.

The specific aims are to:

1. Develop a computer support system to deliver peer-driven, patient-linked Guideline prompts at the point of care using affordable information technology;
2. Evaluate the effect of the Guideline prompt system on the process and outcomes (symptom control, health-related-quality-of-life, ED and hospitalizations) of asthma care; and
3. Evaluate the added effect on outcomes of family-focused, supportive education delivered by a community health worker.

The key product of the computer support system is a guideline prompt that serves as the mechanism for integrating patient specific data with standards of care. 548 children, ages 5-18, with physician diagnosed asthma, enrolled in one Medicaid Managed Care Organization in CT, and receiving care at one of four Federally Qualified Community Health Centers will be recruited. All sites will have access to the computer support system and the to-be-developed, Guideline-Driven Clinical Standards of Asthma Care. In Phase I (12 months), the effect of prompts delivered at the point of care on patient outcomes will be compared to the effect of no-prompt care. In Phase II (6 months), the effect of family-focused, supportive education will be assessed in combination with prompted care compared to no-prompt care and compared to no education. All patients will receive standard screening and outreach to keep appointments. Data will be obtained from medical records, medical and pharmacy claims data as well as patient and parent interviews at baseline and quarterly for 18 months.

ELIGIBILITY:
Inclusion Criteria:

* determined by provider to be asthmatic
* member of Medical Managed Care Organization partner group

Exclusion Criteria:

-

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 548 (Actual)
Dates: Start 2001-08; Primary Completion 2003-05 (Actual); Study Completion 2003-05 (Actual)

PRIMARY OUTCOMES:
asthma control | assessed at all 5 study visits
guideline appropriate medicating by providers | assessed at all 5 study visits
patient knowledge | assessed at all 5 study visits

SECONDARY OUTCOMES:
self efficacy | assessed at all 5 study visits
social support | assessed at all 5 study visits

CONTACTS AND LOCATIONS:
Overall Officials: Judith Fifield, PhD, Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States

REFERENCES:
- [Background] Twiggs JE, Fifield J, Jackson E, Cushman R, Apter A. Treating asthma by the guidelines: developing a medication management information system for use in primary care. Dis Manag. 2004 Fall;7(3):244-60. doi: 10.1089/dis.2004.7.244. PMID 15669584
- [Background] Twiggs JE, Fifield J, Apter AJ, Jackson EA, Cushman RA. Stratifying medical and pharmaceutical administrative claims as a method to identify pediatric asthma patients in a Medicaid managed care organization. J Clin Epidemiol. 2002 Sep;55(9):938-44. doi: 10.1016/s0895-4356(02)00428-6. PMID 12393083
- [Result] Fifield J, McQuillan J, Martin-Peele M, Nazarov V, Apter AJ, Babor T, Burleson J, Cushman R, Hepworth J, Jackson E, Reisine S, Sheehan J, Twiggs J. Improving pediatric asthma control among minority children participating in medicaid: providing practice redesign support to deliver a chronic care model. J Asthma. 2010 Sep;47(7):718-27. doi: 10.3109/02770903.2010.486846. PMID 20812783